CLINICAL TRIAL: NCT06408103
Title: Efficacy of a Multicomponent Intervention on Cognitive Function for the Caregiver-patient Dyad
Acronym: INTERCOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Santander (Other)
Collaborators: Universidad Manuela Beltrán (Other); Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other); Universidad Autónoma de Bucaramanga (Other); Universidad Santo Tomas (Other); Ministerio de Ciencia Tecnología e Innovación - Minciencias (Unknown)
Responsible Party: Principal Investigator, Diana Carolina Tiga, Phd, Epidemiology Ph.D, Universidad de Santander
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTO 652-21
Record Dates: First submitted 2024-04-05; First posted 2024-05-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Rehabilitation; Informal caregiver; Transdisciplinary intervention; Multi-component intervention; Cognitive dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluators responsible for data collection will not have knowledge of the cognitive status or the assignment of participants to study groups. Additionally, the person responsible for subjecting the data to different statistical tests will not be aware of the participants' assignment to the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-component, transdisciplinary and multifocal intervention (intercog-group) (Experimental): This group will receive a multi-component intervention that includes cognitive training, physical exercise, and nutritional counseling; dually and simultaneously. This intervention will be carried out at the patient's home for 12 weeks, with professional support twice a week plus a recommendation to walk 30 minutes/day.
  Furthermore, in the family component, caregivers of the patients will also receive a training component to accompany the intervention and prepare for the caregiver role. This component will be delivered by healthcare professionals in a group format (n=10 per group) over 12 weeks, with weekly sessions lasting 2 hours each. Each session is organized into five parts: opening, activation, education, practice, and explanation of the activities for the next week.
  Interventions: Other: Multi-component, transdisciplinary and multifocal intervention for the cognition
- Usual care plus active control (No Intervention): The conventional management of patients with mild cognitive impairment focuses on therapies such as cognitive rehabilitation, occupational therapy, and physical exercise, with medical monitoring as needed according to the patient's needs. Additionally, they will receive information about infectious diseases such as dengue, pneumonia, tuberculosis, Chagas disease, leishmaniasis, COVID-19, leprosy, urinary tract infection, rabies, superficial and cutaneous mycoses, and hepatitis one topic per week through an infographic and video sent to the cell phone.

INTERVENTIONS:
Other: Multi-component, transdisciplinary and multifocal intervention for the cognition — Multi-component intervention (12 weeks, twice/week, with professional support at home)
  Physical activity for the patient: dual training, strength, balance, with intensity increase monthly, plus moderate walking of 30 minutes/day, 5 days per week.
  Nutritional advice for the patient: Month 1- reduction of added sugars and processed carbohydrates. Month 2- increase consumption of healthy fats and reduction of saturated fats; Month 3- increase in consumption of fruits and vegetables, and a monthly group practical workshop.
  Cognitive training for the patient: activities focused on orientation, attention and concentration, working memory, mathematical reasoning, language, visual construction, executive functions, and reminiscence therapy.
  Accompaniment for the family member: Activities aimed at care and self-care, understanding cognitive deterioration and its progression, support for patient adherence to the intervention, and activities in groups once a week.
  Other Names: INTERCOG
  Arms: Multi-component, transdisciplinary and multifocal intervention (intercog-group)

SUMMARY:
With the aging of the population, an increase in neurocognitive diseases such as dementia is projected. Mild cognitive impairment is considered a precursor stage to dementia, with opportunities for intervention to prevent its progression. Additionally, these illnesses can harm the primary caregiver, who is often an unskilled family member. This is a randomized clinical trial in patients with mild cognitive impairment and their main caregivers.

The intervention will be tested in the dyad for 12 weeks, twice a week with professional support and once a week with caregiver support, the latter will be intervened once a week for 12 weeks. The primary outcome will be the change in cognitive function and its domains. Secondary outcomes will evaluate favorable changes in quality of life in the patient-caregiver couple, frailty, physical capacity, independence, nutritional status, social support, and family caregiver burden. These measurements will be taken at baseline, 3, 6, and 9 months of follow-up. Furthermore, in a subsample of the study population, the taxonomic and metabolomic composition of the intestinal microbiota and the presence of the E4 allele of the APOE (apolipoprotein E) gene will be evaluated before and after the intervention.

DETAILED DESCRIPTION:
Introduction: The aging of the population has led to an increase in the number of individuals with cognitive impairment and neurodegenerative diseases, resulting in greater disability and dependence among older adults worldwide. The prevalence of Mild Cognitive Impairment (MCI) is estimated to be approximately 16%, varying between 2% and 31%.

Multiple interventions have been tested to maintain or improve cognitive function in older adults, including cognitive-motor interventions, yoga, psychosocial and lifestyle interventions, as well as arts-based interventions (dance, theater, music, or visual arts). However, the literature indicates that multicomponent interventions (MCI), also known as multimodal or multidomain, are more effective compared to single-domain interventions in improving cognitive function in older adults.

General Objective: To evaluate the effectiveness of a multicomponent intervention focusing on cognitive function for the caregiver-patient dyad

Methods: Pilot randomized clinical trial, with 1:1 allocation in 102 patients with mild cognitive impairment and their primary caregivers/family members.

Results: The goal is to generate evidence on the efficacy and applicability of these interventions to create a care guide for the caregiver-patient dyad with cognitive impairment, tailored to the Colombian population, with the involvement of different institutions such as universities and healthcare providers.

ELIGIBILITY:
Inclusion and exclusion criteria for elderly adults

Inclusion criteria

1. Age of 55 years or older.
2. Diagnosis of mild cognitive impairment by a Psychiatrist/Neurologist supported by neuropsychological evaluation.
3. Functionality for instrumental activities.
4. Basic proficiency in reading and writing.
5. Absence of untreated hearing impairment and/or uncorrected visual problems.
6. Availability of a primary family caregiver (to be identified).
7. IPAQ with low level of physical activity (pending cutoff point), PARQ and you Fit (pending review).
8. Barthel Index equal to or greater than 80 points.
9. Functional capacity for short-distance ambulation without permanent use of mechanical aids such as wheelchairs.
10. Individuals with a BMI greater than 18.5.
11. Gastrointestinal tract without surgical resections.
12. Tolerance to oral feeding.
13. Vaccination against COVID-19.

Exclusion criteria

1. History of psychosis or congenital intellectual disability.
2. Presence of a central nervous system pathology that could affect cognition (Parkinson's disease, tumors, encephalitis, epilepsy, cerebrovascular disease, traumatic brain injury).
3. Presence of untreated psychiatric disorders, anxiety, depression (Yesavage).
4. Presence of clinically significant systemic diseases (thyroid dysfunction, vitamin B12 deficiency, insulin-dependent diabetes, syphilis, HIV infection, Epstein Barr infection, advanced stage renal failure, cirrhosis). Evaluated through medical history and self-report.
5. Older adult with Chronic Kidney Disease, Hepatopathies (hepatitis, liver cirrhosis),
6. Pulmonary Diseases, or requiring oxygen support, Crohn's Disease, and Colitis.
7. Individual with oncological pathology who has received or is receiving chemotherapy.
8. Individual who has received probiotics or prebiotics in the last 30 days.
9. Presence of clinically significant, active infectious etiology diarrhea.
10. Current or prior abuse of alcohol, tobacco, or drugs.
11. Use of steroids or immunosuppressants in the last 30 days.
12. Recent use of antibiotics, antifungals, or antivirals (excluding topicals) in the last 3 months.
13. Individual who voluntarily decides to withdraw from the study.
14. Older adult without oral, enteral, or parenteral nutritional support.
15. Poor tolerance to exercise, vertigo, medical exercise restriction.

Elimination criteria

1. Institutionalized or hospitalized for more than 1 week, or death during the intervention phase (review and clarity on death).
2. Failure to attend more than 34% of sessions with professional accompaniment (applies to the dyad).

Inclusion and exclusion criteria for caregivers ( Family members)

Inclusion criteria

1. Adults aged 18 years or older.
2. Basic proficiency in reading and writing.
3. Having a level of kinship (consanguineous or non-consanguineous).
4. Vaccination against COVID-19.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in global cognition | 3 months after the intervention, with follow-up at 6 and 9 months
  It will be evaluated by Mini Mental State Examination (MMSE). The scale evaluates the dimensions of orientation, memory, attention and calculation, memory, and language. It has a score of 0 to 30 points and can be categorically interpreted as follows: between 30 and 27 points: No cognitive impairment. Between 26 and 25 points: Possible cognitive impairment. Between 24 and 10 points: mild to moderate cognitive impairment. Between 9 and 6 points: moderate to severe cognitive impairment. Less than 6 points: Major cognitive impairment.
Change in global cognition | 3 months after the intervention, with follow-up at 6 and 9 months
  It will be evaluated by the Montreal Cognitive Assessment (MoCA). The scale evaluates 6 domains: visuospatial ability, executive function, memory, attention/concentration, language, and orientation. It has a scoring scale from 0 to 30, with the following interpretation: 26 or more: No cognitive impairment. 20 to 23: Mild Cognitive Impairment. Score less than 10: major neurocognitive disorder
Change in verbal learning and memory | 3 months after the intervention, with follow-up at 6 and 9 months
  The change in verbal learning and memory will be assessed using the Hopkins Verbal Learning Test (HVLT). It consists of 12 words grouped into three semantic categories. In the population aged between 56 and 76 years, the mean total recall is 18.6 with a standard deviation of 4.6, while for delayed recall, the mean is 6.1 with a standard deviation of 2.4
Change in processing speed and visual attention | 3 months after the intervention, with follow-up at 6 and 9 months
  The change in processing speed and visual attention will be evaluated using the Symbol Digit Modalities Test (SDMT). This test assesses two domains: processing speed and sustained attention. In the population aged between 56 and 76 years, the mean score is 27 (12.1)
Change in visual attention, thinking speed, and visuospatial ability | 3 months after the intervention, with follow-up at 6 and 9 months
  The change in visual attention, thinking speed, and visuospatial ability will be evaluated using the Trail Making Test (TMT-Form A, TMT-Form B). Interpreting the results involves comparing completion times of these forms with normative data corresponding to the same age group. For context, the mean completion times for TMT-A and TMT-B in the population aged 56 to 75 years are as follows: 75.8 seconds (with a standard deviation of 22.8 seconds) for TMT-A and 178 seconds (with a standard deviation of 80.7 seconds) for TMT-B.
Change in executive functioning and selective attention | 3 months after the intervention, with follow-up at 6 and 9 months
  The Color and Word Test assesses executive functioning and selective attention, measuring processing speed and the ability to focus on relevant stimuli while discarding distractors. It also examines cognitive control, inhibition and resistance to cognitive interference. The mean scores for 'Word', 'Color', 'Word-Color' and 'Interference' are 77.7 (standard deviation 21.8), 55.5 (standard deviation 16.6), 30.8 (standard deviation 11.6) and -1.4 (standard deviation 9.1) respectively, reflecting the cognitive abilities of the tested group.
Change in perceptual organization and visual memory | 3 months after the intervention, with follow-up at 6 and 9 months
  The change in perceptual organization and visual memory will be assessed through the Rey Complex Figure Test. This test is divided into 18 elements, each of which scores 2 if the execution is correct; if there is a mistake in the placement or tracing of the element, 1 point is awarded, and if both the placement and tracing are incorrect (or the element is absent), 0 points are awarded. Thus, the total possible score varies between 0 and 36. Two sets of scores are obtained: one for immediate copy and another for long-term recall. In the age group of 56 to 76 years, the mean score for the copying task is 27.9 with a standard deviation of 7.4, while for long-term memory, the mean is 13.7, also with a standard deviation of 7.4
Change in verbal fluency and executive functions | 3 months after the intervention, with follow-up at 6 and 9 months
  Change in verbal fluency and executive functions will be assessed through the Semantic and Phonological Verbal Fluency Test. This test evaluates the ability to generate words following specific semantic or phonological criteria. Scores are assigned based on semantic category and the initial letter of words. For the letter "F," the mean is 9.9 with a standard deviation of 4.3; for "A," the mean is 10.1 with a standard deviation of 4.4; and for "S," the mean is 9.6 with a standard deviation of 4.4. In semantic categories, "ANIMALS" has a mean of 15.6 with a standard deviation of 4.5, while "FRUITS" has a mean of 13 with a standard deviation of 3.7. These scores reflect the quantity and variety of words individuals can produce and are indicative of their linguistic ability and executive capacity
Change in comprehension and expression levels | 3 months after the intervention, with follow-up at 6 and 9 months
  The change in the levels of verbal naming and expression will be assessed from the BOSTON Naming Test. In the age group 56 to 76 years, the mean score for the copying task is 42.8 with a standard deviation of 8
change in verbal comprehension | 3 months after the intervention, with follow-up at 6 and 9 months
  TThe Token Test will be used to assess verbal comprehension. This test specifically measures skills related to listening comprehension and the ability to follow instructions.
  As for the cut-off points for the different ages, they are set as follows: 50 to 56 years (31.5-32), 57 to 59 years (32-32.5), 60 to 68 years (32-32.5), 69 to 71 years (31-31.5), 72 to 74 years (31.5-32.5).
Change WAIS III Digit Retention | 3 months after the intervention, with follow-up at 6 and 9 months
  It is designed to evaluate attention and working memory. It consists of a total of 8 items distributed in two trials. This task is divided into two parts: one that requires repeating the numbers in the order in which they are presented (direct order) and another in the reverse order.
  For individuals between 50 and 71 years of age, the cut-off points for correct retention are 4 in the direct order and 3 in the reverse order. These thresholds indicate the minimum number of digits that the individual must remember correctly to be considered within a normal range of functioning in each task modality

SECONDARY OUTCOMES:
Change in patient independence | 3 months after the intervention, with follow-up at 6 and 9 months
  The patient's independence will be assessed using the Lawton and Brody scale. This scale evaluates functional capacity with 8 items: "ability to use the telephone, shop, prepare food, take care of the house, wash clothes, use transportation, and responsibility regarding medication and administration of their finances." Each item is rated between 0 (dependent) and 1 (independent), and the total score ranges from 0 to 8, reflecting the time required to perform these activities.
Change in physical frailty | 3 months after the intervention, with follow-up at 6 and 9 months
  It will be evaluated using the Linda Fried Frailty Scale, four criteria will be taken: poor physical activity, self-report of physical fatigue, unintentional weight loss, and muscle weakness (estimated by grip strength). The results are interpreted as follows: No criteria = robust, 1 or 2 criteria = pre-frail, 3 or more criteria = frail
Change in nutritional status | 3 months after the intervention, with follow-up at 6 and 9 months
  The nutritional status will be assessed through the Mini Nutritional Assessment (MNA) scale. This scale includes six items: loss of appetite, recent weight loss, mobility, presence of acute illness or psychological stress in the last three months, presence of neuropsychological problems, and body mass index. A score between 12-14 points indicates normal nutritional status, 8-11 points signify a risk of malnutrition, and 0-7 points indicate malnutrition. For a more detailed assessment, three additional items will be evaluated, including whether the patient lives independently, takes more than 3 medications per day, and has skin injuries, through a dichotomous scale of Yes or No
Change in mobility and balance | 3 months after the intervention, with follow-up at 6 and 9 months
  It will be evaluated with the Tinetti Scale. This scale consists of 2 dimensions: mobility and balance, distributed in 9 items. A score of less than 19 points in both dimensions will imply a high risk of falls, a score of 19 to 24 will reflect a medium risk of falls and a score of 25 to 28 will indicate a low risk of falls
Changes in functional capacity and physical condition | 3 months after the intervention, with follow-up at 6 and 9 months
  The assessment will be conducted using the Senior Fitness Test, which consists of six tests grouped into five categories: muscular strength, flexibility, aerobic capacity, agility, and balance.
  Muscular strength is evaluated with two tests: the chair stand test and the arm curl test. Flexibility is assessed using the chair sit-and-reach test and the back scratch test. Aerobic capacity can be evaluated with either the 6-minute walk test or the 2-minute step test. Agility and balance are assessed with the up-and-go test.
  The test scores depend on the participant's gender and age.
Change in the composition of the microbiome | 3 months after the intervention
  Changes in bacterial communities and their metabolites will be assessed using 16S rRNA sequencing for microbiota analysis and both targeted and non-targeted metabolomic approaches for metabolite profiling in blood and stool samples, using mass spectrometry as an analytical technique. This test will be performed on a random sample of patients.
Change in family caregiver overload | 3 months after the intervention, with follow-up at 6 and 9 months
  The caregiver overload is assessed through the Zarit Burden Interview-ZBI, which analyzes the subjective experience of the burden perceived by the caregiver. The scale includes 22 items, scored on a Likert scale of frequency ranging from 1 to 5 points. The total score on the scale can range from 22 to 110 points, with the following categorization: < 46 points: No overload, 46 to 56 points: Mild overload, 57 or more points: Intense overload.
Change in Social Support for Family Caregiver | 3 months after the intervention, with follow-up at 6 and 9 months
  Social support will be determined using the Medical outcomes study social support survey (MOS-SSS). This instrument includes 20 items organized into 4 dimensions: Emotional support, instrumental support, positive social interaction, and affective support. It utilizes a 5-point Likert scale. All items are rated on a 5-point Likert frequency scale. The total score for the global social support index can range from 19 to 95 points, with the following categories: Maximum 95 points, medium 57 points, and minimum 19 points. Low overall social support: <57 points.
Change in quality of life in the dyad | 3 months after the intervention, with follow-up at 6 and 9 months
  Quality of life will be measured through the SF-36 questionnaire applied to the dyad. It consists of 36 questions, in 8 dimensions: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health of the patient. The score is transformed into a scale with a range from 0 (worst health status) to 100 (best health status) and a summary calculation of two dimensions (physical and mental) using the weighted sum of the scores of the eight dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Tiga Loza, Study Director — Universidad de Santander
Locations (1):
- Universidad de Santander / Universidad Manuela Beltrán /FOSCAL, Bucaramanga, Santander Department, Colombia